CLINICAL TRIAL: NCT00958763
Title: Alcohol Use Reduction in Methadone Individuals With HCV
Brief Title: Alcohol Use Reduction in Methadone Individuals With Hepatitis C Virus(HCV)
Acronym: NIAAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Adeline Nyamathi, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G051003101
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Hepatitis C
Keywords: HCV; Alcohol; Methadone Maintained
MeSH Terms: conditions — Hepatitis C | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Motivational Interviewing, Single - MIS (Experimental)
  Interventions: Behavioral: Motivational Interviewing, Single - MIS
- Motivational Interviewing, Group - MIG (Experimental)
  Interventions: Behavioral: Motivational Interviewing Group
- Usual Care Group - UCG (Other)
  Interventions: Other: Usual Care Group - UCG

INTERVENTIONS:
Behavioral: Motivational Interviewing, Single - MIS — The Motivational Interviewing Single Arm is delivered individually to participants in 3 separate sessions to address a specific concept (alcohol use, cravings and what to do with them, and concomitant behaviors and/or consequences of alcohol use). Participants will be encouraged to explore the pros and cons for each of these topics with the facilitator, who will remain non-judgmental. Participants who are eligible for the Hepatitis A/B vaccine are also offered the vaccine in conjunction with each session.
  Other Names: MIS
  Arms: Motivational Interviewing, Single - MIS
Behavioral: Motivational Interviewing Group — The Motivational Interviewing Group Arm is delivered to participants in groups in 3 separate sessions to address a specific concept (alcohol use, cravings and what to do with them, and concomitant behaviors and/or consequences of alcohol use). Participants will be encouraged to explore the pros and cons for each of these topics with the facilitator and with the group, who will remain non-judgmental. Participants who are eligible for the Hepatitis A/B vaccine are also offered the vaccine in conjunction with each session.
  Other Names: MIG
  Arms: Motivational Interviewing, Group - MIG
Other: Usual Care Group - UCG — The Usual Care Arm is delivered to participants in three brief time-equivalent health promotion sessions. Each session focuses on health promoting activities such as the importance of diet and exercise, need for physical and mental health assessment and enhanced coping for those afflicted with a history of drug and alcohol addiction. In addition participants receive liver health promotion education. Participants are also provided referrals to alcohol treatment programs in the community and offered the 3 series hepatitis A/B vaccine
  Other Names: UCG
  Arms: Usual Care Group - UCG

SUMMARY:
The Alcohol Use Reduction in Methadone Individuals with HCV was designed to compare three different types of programs for methadone maintained men and women to determine which of the three programs is most effective for:1) reducing alcohol consumption; 2) improving knowledge of and attitudes toward the disease of hepatitis and the treatment of hepatitis; 3) improving willingness to seek medical care for hepatitis C; 4) completing the 3 sessions on alcohol use reduction; 5) completing the 3 session Hepatitis A and B vaccine; and 6) determining the number of self-reported 12 step alcohol treatment program sessions attended.

DETAILED DESCRIPTION:
Nationwide, major strides have been made in treatment for HCV-infected patients using pegylated interferon and ribaviron; however use of these medications with HCV-infected opioid maintained (OM) IDUs in methadone maintenance (MM) treatment is problematic. Further, as many HCV-infected OM clients are continuing to drink alcohol, ongoing liver fibrosis and other social and behavioral consequences of alcohol use and abuse continue. Despite the fact that brief Motivational Interviewing (MI) has demonstrated effectiveness, these programs are not conducted in MM treatment settings. Moreover, the effectiveness of group delivery, as opposed to one-on-one delivery, of MI is unknown in terms of alcohol use reduction. In Phase I of this two-phased exploratory R21, a qualitative assessment will be conducted with 40 OM HCV-infected adults, 20 moderate alcohol users and 20 heavy alcohol users, equally divided by gender and readiness to change alcohol use, to explore with these clients: 1) factors impacting access to alcohol use reduction and health promotion services and free vaccination for HAV/HBV; and 2) strategies that MM staff can use to assist their clients in seeking services. Staff of a MM clinic will also explore the feasibility of providing these services. In Phase II, we plan to pilot an alcohol use reduction and liver health promotion intervention with 250 eligible, HCV-infected, alcohol-using OM clients receiving MM. Two intervention groups incorporating MI) will provide on-site brief MI (3 sessions) counseling to participants using either one-on-one delivery (MI-Single) or the group-delivery (MI-Group). In addition, each group will be offered the Liver Health Promotion (LHP) program, which includes a 30-minute health promotion education session, referral to a community 12-Step alcohol outpatient program, and an offer for free screening for HAV/HBV, and the HAV/HBV vaccination series, if eligible (defined as being HAV and/or HBV seronegative). All these services will be integrated within participants' usual MM clinic onsite services. A third group, the Usual Care (UC) group will receive the same components offered to the intervention groups except for a time balanced on-site brief 3 session health promotion counseling as opposed to the MI. The short-term goals of the proposed study are to refine strategies that can be fully tested in a large-scale intervention trial. The long-term goals are to contribute to knowledge about promoting alcohol-related health-seeking and treatment completion behaviors in MM clinic settings that serve OM HCV-positive clients, so that population-specific intervention strategies can be developed.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be 18 - 55 years of age, enrolled at the participating methadone maintenance clinic for the past 2 months, and moderate to heavy alcohol users within the last 3 months

Exclusion Criteria:

* Individuals who are not within the age range, have not been enrolled in a methadone maintenance clinic for the past 2 months and were not moderate to heavy alcohol users within the last 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 219 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Compare two Motivational Interviewing (MI) groups with the Usual Care group at six-month follow-up on reduction of alcohol use, and determine whether group MI delivery is as effective as individual MI delivery in relation to decreased alcohol use | 2 years

SECONDARY OUTCOMES:
Determine whether there are differential rates of attendance in the programs, and, for eligible participants, contrast the three groups on completion of the HAV/HBV vaccination series, and number of self-reported visits to 12-step alcohol programs. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Nyamathi, PhD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - Matrix Institute, Los Angeles, California
  - Bay Area Addiction Research & Treatment, Inc (BAART), Los Angeles, California
  - Tri-City Institute, Los Angeles, California